CLINICAL TRIAL: NCT05591989
Title: Clinical Evaluation of Safety and Efficacy for the NEUROMARK System in Subjects With Chronic Rhinitis (PARAGON) - A Prospective, Single-arm, Multicenter Clinical Study.
Brief Title: Clinical Evaluation of Safety and Efficacy for the NEUROMARK System in Subjects With Chronic Rhinitis (PARAGON)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurent Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0007
Record Dates: First submitted 2022-10-18; First posted 2022-10-24 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Chronic Rhinitis
Keywords: Rhinitis
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Intervention Model Description: A prospective, single-arm, multicenter clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Subjects will undergo treatment with the NEUROMARK System
  Interventions: Device: NEUROMARK System

INTERVENTIONS:
Device: NEUROMARK System — The NEUROMARK System is indicated for use in otorhinolaryngology (ENT) surgery for creation of radiofrequency (RF) lesions to disrupt posterior nasal nerves in patients with chronic rhinitis.

SUMMARY:
The PARAGON Study is a prospective, single-arm, multicenter safety and efficacy study of the Neurent Medical NEUROMARK System in subjects with chronic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

Subjects MUST:

1. Be ≥18 years of age.
2. Have been experiencing rhinitis symptoms for a minimum of 6 months.
3. Have moderate to severe symptoms of runny nose (individual rTNSS symptom rating of 2 or 3), mild to severe symptoms of nasal congestion (individual rTNSS symptom rating of 1,2, or 3), and a minimum total score of 5 (out of 12) at baseline.
4. Have an allergy test (by skin prick or intradermal testing, or by a validated in vitroImmunoglobin E [IgE test]) on file within 5 years of the baseline visit or is willing to have one performed during the study prior to 6-month visit.
5. Be an appropriate candidate for bilateral NEUROMARK® device treatment performed under local anesthesia.
6. Test negative for active COVID-19 at the start of the study screening and continue to be free of COVID-19 symptoms until the time of enrollment/treatment.
7. Be willing and able to comply with all study elements, as indicated by written informed consent.

Exclusion Criteria:

Subjects MUST NOT:

1. Have clinically significant anatomic obstruction that in the investigator's opinion limit access to the posterior nose, including but not limited to severe septal deviation or perforation, nasal polyps, and/or sinonasal tumor.
2. Have had previous sinus or nasal surgery within 6 months of study enrollment.
3. Have previously undergone RF, cryotherapy, or other surgical interventions for rhinitis.
4. Have an active nasal or sinus infection.
5. Have nasal mucosal erosion/ulceration.
6. Have rhinitis symptoms that are due to seasonal allergies only.
7. Have plans to (or otherwise anticipates the need to) undergo an ENT procedure concurrently or within 6 months after the study procedure.
8. Have started a new sinonasal medication regimen within 4 weeks prior to treatment that, according to the manufacturer's labelling, has not yet stabilized.
9. Be on prescribed anticoagulants (eg, warfarin, Plavix) or ≥ 325 mg aspirin that cannot be held for an appropriate time before the procedure.
10. Have a history of chronic epistaxis or experienced a significant epistaxis event (defined as epistaxis requiring medical intervention) in the past 3 months.
11. Have numbness of the soft palate, excessive dry eye, excessive dry nose, or other indication of neuro/nerve compromise in the sinonasal cavity.
12. Have an active rhinitis medicamentosa or a history of rhinitis medicamentosa within the past 6 months.
13. Have been diagnosed with atrophic rhinitis.
14. Have had previous head and/or neck irradiation.
15. Have an allergy or intolerance to local anesthetic agents.
16. Be pregnant.
17. Have a physical, neurological, medical, psychiatric condition or situation that, in the investigator's opinion, puts the subject at risk, could confound the study results, or may interfere significantly with the subject's participation in the study.
18. Be participating in another clinical research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Safety | 24 months
  Safety, as assessed by the incidence of device- and/or procedure related serious adverse events (SAEs)
Efficacy | 6 months
  Efficacy, as assessed by the mean change from baseline in nasal symptoms using the 4-symptom rTNSS (reflective Total Nasal Symptom Score) at 6-month follow-up (FU)

SECONDARY OUTCOMES:
The mean change from baseline in rTNSS total score (except 6-month FU) | 24 months
  The mean change from baseline in rTNSS total score (except 6-month FU)
The mean change from baseline in rTNSS subscores | 24 months
  The mean change from baseline in rTNSS subscores
The mean change from baseline in Mini Rhinoconjunctivitis Quality of Life Questionnaire (mini-RQLQ) score | 24 months
  The mean change from baseline in Mini Rhinoconjunctivitis Quality of Life Questionnaire (mini-RQLQ) score
The mean change from baseline in Clinical Global Impression -Improvement (CGI-I) score | 24 months
  The mean change from baseline in Clinical Global Impression -Improvement (CGI-I) score
Percent of subject satisfaction at follow-up | 24 months
  Percent of subject satisfaction at follow-up
Tolerability of treatment via verbal report using the Numeric Rating Scale (NRS) score | 24 months
  Tolerability of treatment via verbal report using the Numeric Rating Scale (NRS) score

CONTACTS AND LOCATIONS:
Overall Officials: Annalise Sorensen, Study Director — Neurent Medical
Locations (10):
- United States (10):
  - Alabama Nasal and Sinus Center (Alabama Allergy), Birmingham, Alabama
  - Sacramento ENT, California City, California
  - United Medical Doctors, Temecula, California
  - Colorado ENT, Colorado Springs, Colorado
  - New Orleans Sinus Center, Marrero, Louisiana
  - Centers for Advanced ENT Care (CAdENT), Baltimore, Maryland
  - Rontal Clinics, Royal Oak, Michigan
  - Specialty Physician Associates, Bethlehem, Pennsylvania
  - Richmond ENT, Richmond, Virginia
  - Ear Nose Throat & Allergy Associates, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yen DM, Davis GE, Ow RA, O'Malley EM, Del Signore AG. Two-Year Clinical Outcomes After Multipoint Impedance-Controlled Radiofrequency Ablation of the Posterior Nasal Nerve for Treatment of Chronic Rhinitis. Ear Nose Throat J. 2025 Oct 9:1455613251382759. doi: 10.1177/01455613251382759. Online ahead of print. PMID 41065547
- [Derived] Davis GE, Ow RA, Yen DM, O'Malley EM, Del Signore AG. Clinical Outcomes After Innovative Multipoint Impedance-Controlled Radiofrequency Ablation of the Posterior Nasal Nerve for Treatment of Chronic Rhinitis. Ear Nose Throat J. 2024 Sep 24:1455613241285134. doi: 10.1177/01455613241285134. Online ahead of print. PMID 39315465